CLINICAL TRIAL: NCT07138677
Title: The Safty and Efficacy of Mild Cognitiive Impairment Network Guided Transcranial Magnetic Stimulations for Patients With Early Alzheimer's Disease (SENS-eAD): A Randomized, Double-blind Trial
Brief Title: Safty and Efficacy of MCI Network Guided TMS for Early Alzheimer's Disease: A Randomized, Double-blind Trial
Acronym: SENS-eAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Director of medical psychological department, Anhui Medical University, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AHMU-NetTMS-eAD
Record Dates: First submitted 2025-04-30; First posted 2025-08-24 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer's Disease; Transcranial Magnetic Stimulation; Individualized Navigation
Keywords: Alzheimer's Disease; Transcranial Magnetic Stimulation; Individualized navigation
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MCI real group (Experimental): Stimulation delivered by a real coil through MagStim Rapid2 and guided by BrainSight navigation system.
  Interventions: Other: transcranial magnetic stimulation
- MCI sham group (Sham Comparator): Stimulation delivered by a sham coil through MagStim Rapid2 and guided by BrainSight navigation system.
  Interventions: Other: transcranial magnetic stimulation

INTERVENTIONS:
Other: transcranial magnetic stimulation — Neuronavigated Theta-Burst Transcranial Magnetic Stimulation

SUMMARY:
Estimate the safty and efficacy of personalized network neuronavigated transcranial magnetic stimulations in early Alzheimer's disease patients

DETAILED DESCRIPTION:
All patients undergo a series of medical assessments that include physical examination and routine laboratory studies before and after repetitive transcranial magnetic stimulation (rTMS) treatment. Upon meeting the inclusion criteria and providing informed consent, each participant will complete a series of cognitive assessments and rTMS treatments at the First Affiliated Hospital of AnHui medical university. Stratified block randomization will be used to assign participants to different intervention groups. Stratification is based on Mini-Mental State Examination (MMSE) scores (<24 vs. ≥24), and randomization will be conducted using variable block sizes of 4 or 6.

For each participant, the investigators will compute their persoanlized dorsal prefrontal targets by using their own resting-state functional MRI data and a predefined MCI network. They will then be randomly assigned to receive real or sham rTMS treatment for two weeks. The sham stimulations will be delivered by a sham coil. All the experiment procedures are the same between groups except the coil.

With a statistical power of 0.8, an effect size of 0.96, a significance level of 0.05, and a 5% expected dropout rate, the final sample size is 20 participants per group. In this double-blind study, patients and clinical raters are masked to the allocated conditions. Only one investigator responsible for group allocation has access to the randomization list.

Each participant will be treated for 14 days by rTMS. Before the rTMS treatment, a trained investigator will perform a series of cognitive assessments and neuropsychological tests. The ADAS-Cog is the primary outcome. Other tasks and questionnaires include cognition (including MoCA, MMSE, DS, Stroop test, BNT-30, VFT, CDT, JLOT. Form H, HVOT), memory (CAVLT, LMT), emotion (HAMA-17,HAMD-14), behavioral and psychological symptoms (NPI), and treatment tolerability. All the tests will be conducted within two days. The participants undergo a multi-modal MRI scan and an electroencephalogram (EEG) examination.

The participants also undergo the ADAS-cog, a battery of neuropsychological tests, multi-modal MRI, and EEG examinations. participants will be instructed to focus their answers on the past 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subject diagnosed as either mild cognitive impairment due to AD or mild AD dementia based on National Institute on Aging-Alzheimer's Association criteria.
2. MMSE score 18-28.
3. CDR score 0.5-1.
4. On stable treatment with IAChE or memantine for at least 6 months.
5. Literate in Han Chinese.

Exclusion Criteria:

1. Recevied rTMS treatment in the past 3 months.
2. Depression or other psychiatric disorders.
3. History of head injury, stroke, epilepsy or other neurologic disease.
4. Organic brain defects on T1 or T2 images.
5. History of unexplained loss of consciousness.
6. Implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, or any implanted medical device that is incompatible with MRI.
7. Family history of medication refractory epilepsy.
8. History of substance abuse within the last 6 months.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Alzheimers Disease Assessment Scale Cognitive section (ADAS-Cog) | Baseline and 2 weeks
  The changes in Alzheimers Disease Assessment Scale Cognitive section (ADAS-Cog) will constitute the major research outcome measure used to assess response to transcranial magnetic stimulation (TMS). The ADAS-COG scale tests orientation, language, structure, use of ideas, immediate recall of words and word re-recognition, and consists of 11 questions out of a possible 70 points, with the higher the score the more cognitively impaired.

SECONDARY OUTCOMES:
Mini Mental State Examination (MMSE) | Baseline and 2 weeks
  The changes in MMSE will constitute the primary research outcome. The full name of MMSE is mini-mental state examination, and the scale consists of 30 subject, include the following seven aspects: time orientation, place orientation, immediate memory, attention and calculation, delay memory, language, visual space. One point is awarded for each question correctly answered during MMSE evaluation. If subject give the wrong answer or don't know answer he/she awarded 0 score, scope of scale score of 0 to 30 points. The higher the score, the better. In this study, changes in MMSE scores before and after treatment were used as secondary outcome measure.
Montreal Cognitive Assessment (MoCA) | Baseline and 2 weeks
  The changes in MoCA will be used to assess the response to TMS. MoCA was developed by Nasreddine et al. based on clinical experience and reference to the MMSE cognitive items and scores, and the final version was finalized in November 2004. The investigators adopted a localized version (Mandarin version#includes 2 alternative versions) in line with the Chinese cultural background. It includes 11 inspection items in 8 cognitive fields, including visual structure skills, executive function, naming, attention and calculation, language, abstract thinking, memory, and orientation. The normal score range from 26 to 30. Anyone who has been education for less than 12 years will need to add one point to his final score. The final score of the higher the better.
Digital Span Test; Forward and Backward (DST) | Baseline and 2 weeks
  The changes in DST will constitute the secondary research outcome. Digital span test (DST) was commonly used to evaluate attention ability and instantaneous memory ability. There are two types of test: forward (0-14) and backward (0-13). In the forward test, the subjects were asked to retell the the digits immediately after hearing it untilthey could not be repeated correctly. In backward test, the subjects were asked to repeat a set of numbers in reverse order until they could not be repeated correctly. The length of the last set of Numbers correctly repeated by the subjects was the final score, forward and backward are counted separately. The higher the score, the better.
Hamilton Depression Scale (HAMD) | Baseline and 2 weeks
  Hamilton Depression Scale (HAMD) compiled by Hamilton in 1960, is the most common clinical to assess Depression Scale. In this study, we selected the HAMD version with 17 questions. Subjects were assessed for their depression in the past week. Each question scored between 0 and 4 points. Higher scores indicate more depressive symptoms. The severity of the disease and the therapeutic effect can be evaluated after treatment.
Hamilton Anxiety Scale (HAMA) | Baseline and 2 weeks
  Hamilton Anxiety Scale (HAMA) was compiled by Hamilton in 1959. It was one of the most commonly used scales in psychiatric clinic, including 14 items. It is often used in clinical diagnosis and degree classification of anxiety disorder. The subjects were assessed for their anxiety in the past week. Each question scored between 0 and 4 points. The higher the score, the more symptoms of anxiety.
Neuropsychiatric Inventory (NPI) | Baseline and 2 weeks
  The Neuropsychology Scale (NPI) evaluates 12 neuropsychiatric disorders which included 10 neuropsychiatric symptoms and 2 autonomic neurological symptoms based on the caregiver's perception of the patient's behavior and the perceived distress. Each item was evaluated for its occurrence frequency (1-4 points) and severity (1-3 points). The frequency and severity were multiplied to obtain the score (0-12 points) of each item.The patient's assessment rating ranges from 0 to 144, and the caregiver's distress rating score is 0 to 60. The lower the score, the lighter the symptoms.
Judgment of line Judgment of line orientation test (JLOT) | Baseline and 2 weeks
  The JLOT test was determined by Benton et al. in 1994. There are two versions of H and V. The difference is that the order in which the pictures are presented is different. Each version contains 35 images, of which the official test consists of 30 images, and the other 5 images are for the participants to learn. The final score is the correct number of subjects to answer, the full score is 30 points, the higher the score, the better the space perception ability of the subject.
Hooper visual organization test (HVOT) | Baseline and 2 weeks
  HVOT is a cognitive test used to evaluate the perceived structure of the subject. It consists of 30 items (1 point each question) and the total score is 30 points. The final score is the correct number of subjects to answer, the full score is 30 points. The higher the score, the better the space perception ability of the subject.
The Stroop color word test | Baseline and 2 weeks
  The Stroop color word test was developed by Stroop in 1935 and is used to evaluate the attention function of the subject. The subject is required to correctly read the target color on the stimulus card and record the completion time. The final completion time is the score of the participant. The shorter the time used, the better the performance of the subjects.
EEG | Baseline and 2 weeks
  EEG data were obtained from each subject based on 64 electrode locations of the International 10-20 system (sampling frequency 1000Hz).
Logic Memory Test (LMT) | Baseline and 2 weeks
  The Logical Memory test, part of the Wechsler Memory Scale, primarily assesses an individual's verbal memory capabilities. The test involves presenting two brief stories to the subject, who is then asked to immediately recall and subsequently recall them after a delay. By comparing the immediate and delayed recall performance, the subtest evaluates both short-term and long-term memory retention.
Pittsburgh Sleep Quality Index (PSQI) | Baseline and 2 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a standardized tool used to assess individual sleep quality. It consists of 19 self-rated items that evaluate sleep quality, covering 7 aspects including sleep duration, efficiency, disturbances, and others. Each component is scored from 0 to 3, with higher scores indicating poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No